CLINICAL TRIAL: NCT06148532
Title: EnCoRe MoMS Aim 2: Engaging Communities to Reduce Morbidity From Maternal Sepsis
Brief Title: EnCoRe MoMS: Engaging Communities to Reduce Morbidity From Maternal Sepsis (Aim 2)
Status: Enrolling by invitation | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Northern Manhattan Perinatal Partnership (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dena Goffman, Ellen Jacobson Levine and Eugene Jacobson Professor of Women's Health (in Obstetrics and Gynecology), Columbia University
Other Study IDs: AAAU3697 - Aim 2; 1UG3HD111247 (NIH)
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Maternal Sepsis; Infections
Keywords: Electronic Health Record; Post Partum Period; Pregnancy; Maternal Health
MeSH Terms: conditions — Pregnancy Complications, Infectious; Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PRC Database: EHR records for hospital delivery admissions and postpartum readmissions obtained from Perinatal Research Consortium (PRC) sites to be harmonized with SDoH data and analyze to optimize sepsis risk prediction.

SUMMARY:
Sepsis is the second leading cause of maternal death in the U.S. For racial and ethnic minoritized birthing people, especially those who are Black, living in poverty, and from underserved communities, labor and postpartum are particularly vulnerable risk periods. The goal of this multi-center, multidisciplinary observational study is to optimize risk prediction accounting for the social determinants of health, and establish a novel maternal care continuity model to reduce sepsis- related death and disability and increase maternal health equity.

DETAILED DESCRIPTION:
Maternal sepsis is the second leading cause of maternal death, major cause of morbidity, and preventable in most cases. EnCoRe MoMS: Engaging Communities to Reduce Morbidity from Maternal Sepsis will (Aim 2) Develop algorithms to optimize prediction of sepsis around delivery and postpartum.

In the UG3 phase, robust community engagement and research infrastructures were established to: Aim 2a. Create a rich electronic health records (EHR) database from the Perinatal Research Consortium (PRC). Aim 2b. Collate neighborhood-level datasets characterizing social determinants of health (SDOH)

In the UH3 phase, the investigators will Aim 2c. Harmonize patient-level EHR and neighborhood-level SDOH datasets and use machine learning models to analyze the individual and joint contributions of patient and neighborhood factors to optimize sepsis risk prediction within the PRC sample.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Delivery admission (and) postpartum readmission at one of the Perinatal Research Consortium sites 2014-2021

Exclusion Criteria:

* Under 18 years old
* Delivery admission (and) postpartum readmission at hospital that is not in the Perinatal Research Consortium
* Delivery admission before 2014 or after 2021

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Delivery admission records at PRC sites
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Maternal sepsis risk | Delivery hospitalization through 8 weeks postpartum
  Sepsis as evaluated by the following scoring systems: Sepsis-2 (proven or suspected infection in combination with at least two systemic inflammatory response syndrome criteria); Sepsis-3 (organ dysfunction as defined by an acute change in total organ dysfunction score within 24 hours of suspected infection); and Center for Disease Control (CDC) Sepsis (presumed infection and organ dysfunction based on CDC criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Dena Goffman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia Unviersity Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No